CLINICAL TRIAL: NCT01106339
Title: Phase 1 Study of Immune, Psychometric and Sociodemographic Patterns in Pain Patients Classified by DSM-IV
Brief Title: Immune Patterns in Pain Patients DSM-IV
Acronym: IPPPDIV
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: University Hospital Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, MBA, University of Ulm
Other Study IDs: Anae_Pain_Ulm_DSM-IV
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Somatoform Disorders; Fibromyalgia; Myofascial Pain Syndrome, Diffuse; Depression; Chronic Fatigue Syndrome
Keywords: humans; patients; somatoform disorders; fibromyalgia; myofascial pain syndrome diffuse; depression; chronic fatigue syndrome; inflammation; inflammatory response; biomarkers; cytokines; cell surface markers; functional polymorphisms
MeSH Terms: conditions — Somatoform Disorders; Fibromyalgia; Depression; Fatigue Syndrome, Chronic; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, and white cells will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients with somatoform disorders due to DSM-IV

SUMMARY:
The purpose of this study is to define subgroups of patients with somatoform disorders due to DSM-IV by immunological, psychological and genetic characterization.

DETAILED DESCRIPTION:
Pain patients are defined as patients with a somatoform disorder due to DSM-IV, if chronic pain lasts for at least 6 months in several anatomical regions. Somatoform disorders (DSM-IV) have the presence of physical symptoms that suggest a general medical condition but that are not fully explained by a general medical condition, by the direct effects of a substance, or by another mental disorder. The symptoms must cause clinically significant distress or impairment in social, occupational, or other areas of functioning. The physical symptoms are not under voluntary control. Psychic factors exclusively or in combination with a medical disease factor influence onset, severity, exacerbation or maintenance of symptoms decisively. A subgroup of somatoform disorders, i.e., fibromyalgia, is a common nonarticular rheumatic syndrome characterized by myalgia and multiple points of focal muscle tenderness to palpation (trigger points). Muscle pain is typically aggravated by inactivity or exposure to cold. This condition is often associated with general symptoms, such as sleep disturbances, fatigue, stiffness, headaches, and occasionally depression. There is significant overlap between fibromyalgia and the chronic fatigue syndrome. Fibromyalgia may arise as a primary or secondary disease process. Interleukins IL-1ß, IL-6 und tumor necrosis factor-a have been detected in the skin of these patients. Blockade of the 5HT3 receptor has been reported to alleviate chronic pain in tendopathy, fibromyalgia and autoimmune diseases. However, only a subgroup of patients responds to this therapy. It is supposed that patients with somatoform disorders (DSM-IV) diagnosed according to clinical criteria consist of immunologically heterogenous groups. However, up to now, the immunologic and genetic background of patients with somatoform disorders classified via DSM-IV has not been systematically evaluated. The study concentrates on the psychometric characterization of patients with pain disorder focusing on depression, anxiety, coping behavior, psychic trauma, alexithymia and somatoform symptoms. The present study is performed to define subgroups of patients with somatoform disorders (DSM-IV) by immunological, pyschologic and genetic characterization which may benefit from potential 5HT3 receptor antagonists or anti-inflammatory therapy.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain patients with a somatoform disorder due to DSM-IV
* chronic pain > 6 months in several anatomical regions
* presence of physical symptoms that suggest a general medical condition
* the symptoms must cause clinically significant distress or impairment in social, occupational, or other areas of functioning
* the physical symptoms are not under voluntary control
* Psychic factors exclusively or in combination with a medical disease factor influence onset, severity, exacerbation or maintenance of symptoms decisively
* fibromyalgia

Exclusion Criteria:

* age < 18 years
* psychosis
* symptoms fully explained by a general medical condition, by the direct effects of a substance, or by another mental disorder
* pregnancy
* inclusion in other studies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic pain patients with a somatoform disorder due to DSM-IV
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pattern of inflammatory biomarkers | 1 year

SECONDARY OUTCOMES:
Pattern of cell surface markers | 1 year
Functional polymorphisms | 1 year
Psychometric tests | 1 year
Demographic tests | 1 year
Severity of pain | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Steffen, MD, Principal Investigator — Clinic of Anesthesiology, University Hospital Medical School, Steinhoevelstrasse 9, 89070 Ulm, Germany
Locations (1):
- Clinic of Anesthesiology, Dept. of Pain, Ulm, Germany

REFERENCES:
- [Background] Schneider EM, Ma X, Stratz T, Muller W, Lorenz I, Seeling WD. Immunomodulatory function of the 5-HT3 receptor antagonist tropisetron. Scand J Rheumatol Suppl. 2004;119:34-40. PMID 15515411